CLINICAL TRIAL: NCT00880542
Title: A Phase II Study of Sorafenib and Ifosfamide as a Treatment for Patients With Sarcoma
Brief Title: Sorafenib and Ifosfamide in Treating Patients With High-Grade Soft Tissue Sarcoma or Bone Sarcoma That Can Be Removed by Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study lost funding.
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000633030; UCLA-0704086; BAYER-UCLA-0704086; ONYX-UCLA-0704086
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Results first posted 2011-05-10 (Estimated); Last update posted 2020-08-10 (Actual); Status verified 2012-07

CONDITIONS: Sarcoma
Keywords: localized osteosarcoma; stage II adult soft tissue sarcoma; stage III adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Sorafenib; Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib + Ifosfamide (Experimental): * Neoadjuvant therapy: Patients receive oral sorafenib tosylate twice daily on days 1-14 in course 1. Patients then receive oral sorafenib tosylate twice daily on days 1-28 and ifosfamide IV continuously on days 1-7 in courses 2 and 3. Treatment repeats every 14-28 days* for 3 courses.
  NOTE: *Course 1 is 14 days in duration; courses 2 and 3 are 28 days in duration.
  * Surgery: At least 1 week after the completion of neoadjuvant therapy, patients undergo surgery.
  * Adjuvant therapy: Beginning ≥ 3 weeks after surgery, patients who respond to neoadjuvant therapy receive oral sorafenib twice daily for 6 months. Patients also receive 2 courses of ifosfamide as in courses 2 and 3 of neoadjuvant therapy.
  Interventions: Drug: sorafenib; Drug: Ifosfamide

INTERVENTIONS:
Drug: sorafenib — Patients with sarcoma who have resectable disease will be treated with neoadjuvant sorafenib and ifosfamide. PET/CT will be used to assess the metabolic and radiographic response to therapy.
Drug: Ifosfamide — Patients with sarcoma who have resectable disease will be treated with neoadjuvant ifosfamide and sorafenib. PET/CT will be used to assess the metabolic and radiographic response to therapy.

SUMMARY:
RATIONALE: Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as ifosfamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving sorafenib together with ifosfamide may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects of giving sorafenib together with ifosfamide and to see how well it works in treating patients with high-grade soft tissue sarcoma or bone sarcoma that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the safety, toxicity, and efficacy of neoadjuvant sorafenib tosylate and ifosfamide in patients with resectable high-grade soft tissue or bone sarcoma.

Secondary

* Assess the long-term efficacy or impact of therapy in these patients, in terms of the duration of local recurrence-free survival, distant recurrence-free survival, and disease-specific survival.

OUTLINE:

* Neoadjuvant therapy: Patients receive oral sorafenib tosylate twice daily on days 1-14 in course 1. Patients then receive oral sorafenib tosylate twice daily on days 1-28 and ifosfamide IV continuously on days 1-7 in courses 2 and 3. Treatment repeats every 14-28 days* for 3 courses.

NOTE: *Course 1 is 14 days in duration; courses 2 and 3 are 28 days in duration.

* Surgery: At least 1 week after the completion of neoadjuvant therapy, patients undergo surgery.
* Adjuvant therapy: Beginning ≥ 3 weeks after surgery, patients who respond to neoadjuvant therapy receive oral sorafenib twice daily for 6 months. Patients also receive 2 courses of ifosfamide as in courses 2 and 3 of neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed high grade sarcoma of the soft tissue or bone
* participants Identified as a proper candidate for ifosfamide-based neoadjuvant therapy
* candidates must have operable disease for which a resection is planned
* ECOG performance status 0-1
* Hemoglobin ≥ 9.0 g/dL
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT and AST ≤ 2.5 times ULN (≤ 5 times ULN for patients with liver involvement)
* INR < 1.5 or PT/PTT normal.Concurrent anticoagulation therapy with warfarin or heparin allowed
* Creatinine ≤ 1.5 times ULN
* women of childbearing potential must have negative pregnancy test performed within 7 days prior to start of treatment.
* Fertile patients must use effective contraception during and for ≥ 2 weeks after completion of study therapy.
* A signed informed consent must be obtained prior to any study specific procedures.

Exclusion Criteria:

* known HIV infection
* chronic hepatitis B or C infection
* clinically active serious infection > CTCAE grade 2
* NYHA class III or IV congestive heart failure
* unstable angina (i.e., anginal symptoms at rest) or new onset angina within the past 3 months
* myocardial infarction within the past 6 months
* cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* uncontrolled hypertension (i.e., systolic blood pressure [BP] > 150 mm Hg or diastolic BP > 90 mm Hg) despite optimal medical management
* thrombolic or embolic events (e.g., cerebrovascular accident, including transient ischemic attacks) within the past 6 months
* pulmonary hemorrhage or bleeding event ≥ CTCAE grade 2 within the past 4 weeks
* other hemorrhage or bleeding event ≥ CTCAE grade 3 within the past 4 weeks
* Any condition that would impair the ability to swallow whole pills
* malabsorption problem
* Any known severe hypersensitivity to sorafenib tosylate or any of its excipients
* known or suspected allergy to sorafenib tosylate or any agent given in this study
* serious nonhealing wound, ulcer, or bone fracture
* evidence or history of bleeding diathesis or coagulopathy
* significant traumatic injury within the past 4 weeks
* major surgery or open biopsy within 4 weeks of starting treatment
* Concomitant St. John's wort or rifampin
* KNown brain metastases. Patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastases.
* any condition that impairs patients' ability to swallow pills
* any malabsorption problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-08; Primary Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Tap, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period: 08/20/2008 - 07/19/2010 Types of location: Academic medical clinics
Pre-assignment Details: There are no pre-assignment details to describe
Period: Treatment Period (Sorafenib+Ifosfamide)
Arm/Group | Sorafenib + Ifosfamide
Started | 7
Completed | 4
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — disease progression | 2
Period: Response Evaluation Period(REP): PET/CT
Arm/Group | Sorafenib + Ifosfamide
Started | 4
Completed | 4
Not Completed | 0
Period: REP: Surgical Resection
Arm/Group | Sorafenib + Ifosfamide
Started | 4
Completed | 3
Not Completed | 1
Not completed — progressive disease | 1
Period: Post Surgical Evaluation
Arm/Group | Sorafenib + Ifosfamide
Started | 3
Completed | 3 (none of the 3 subjects met study criteria for continuation of therapy.)
Not Completed | 0
Period: Continued Treatment Period
Arm/Group | Sorafenib + Ifosfamide
Started | 0 (None of the 3 subjects from previous period met study criteria for continuation of therapy.)
Completed | 0
Not Completed | 0
Period: Follow-up Period
Arm/Group | Sorafenib + Ifosfamide
Started | 7 (All 7 patients who started the treatment period completed the follow-up period.)
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib + Ifosfamide
Number analyzed (Participants) | 7
Age, Continuous [Median (Full Range); unit: years] | 56 [33 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Using PET/CT Scan to Measure Safety, Toxicity, and Efficacy of Neoadjuvant Sorafenib Tosylate and Ifosfamide in Patients With Resectable High-grade Soft Tissue or Bone Sarcoma.
Description: After cycle 1, a limited PET/CT scan of the affected site will be performed to assess response to sorafenib treatment alone. After cycle 3, prior to surgery, a limited PET/CT scan of the affected site will be performed to assess response to the combination sorafenib and ifosfamide treatment.
Time Frame: Participants were followed for duration of study, an average of 1 year.
Population: Due to the study closing early and the few number of participants enrolled, the outcome measures were not done.
Arm/Group | Sorafenib + Ifosfamide
Number analyzed (Participants) | 0

2. Secondary Outcome: Local and Distant Recurrence-free Survival
Time Frame: conclusion of study
Population: Due to study closing early and the few number of participants enrolled, the outcome measures were not done.
Arm/Group | Sorafenib + Ifosfamide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event(AE)data collected between 08/20/2008 and 7/19/2010, therefore AE reporting period is approximately 1 year and 11 months.
Description: Systemic adverse event assessment with every physician contact day, either as outpatient or inpatient throughout the active treatment phase of the study and every three months in the follow-up period.
Arm/Group | Sorafenib + Ifosfamide
Serious Adverse Events (participants affected / at risk) | 4/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib + Ifosfamide (N=7)
Grade 3 and 4 Neutropenic fever related to Ifosfamide (Blood and lymphatic system disorders) | 2
Grade 3 lower back pain due to disease or GCSF (Musculoskeletal and connective tissue disorders) | 1
Grade 3 thrombocytopenia related to Ifosfamide (Blood and lymphatic system disorders) | 1
Grade 3 lymphopenia related to Ifosfamide (Blood and lymphatic system disorders) | 1
Grade 3 hypocalcemia related to possible vitamin D insufficiency (Metabolism and nutrition disorders) | 1
Grade 4 bowel perforation due to disease progression (Gastrointestinal disorders) | 1
Grade 4 leukocytopenia related to Ifosfamide (Blood and lymphatic system disorders) | 1
Grade 4 Neutopenia related to Ifosfamide (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib + Ifosfamide (N=7)
Epistaxis (General disorders) | 1
Neutropenia fever (Infections and infestations) | 1
Anemia (Blood and lymphatic system disorders) | 3
Elevated international normalized ratio (INR) (Hepatobiliary disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Tachycardia (Cardiac disorders) | 2
Chest pain (Cardiac disorders) | 1
chills (General disorders) | 1
Fatigue (General disorders) | 2
shaking spells (General disorders) | 1
weight loss (General disorders) | 1
fever (General disorders) | 2
alopecia (Skin and subcutaneous tissue disorders) | 2
anal fissure (Skin and subcutaneous tissue disorders) | 1
bleeding with bowel movement (Skin and subcutaneous tissue disorders) | 1
calluses, finger/toes (Skin and subcutaneous tissue disorders) | 1
desquamation (Skin and subcutaneous tissue disorders) | 1
ecchymosis below left eye (Skin and subcutaneous tissue disorders) | 1
hand-foot syndrome (Skin and subcutaneous tissue disorders) | 1
Lt. heel plantar foot tenderness (Skin and subcutaneous tissue disorders) | 1
Painful blister on hand (Skin and subcutaneous tissue disorders) | 1
Pionidal hidratitis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Purpura right arm (Skin and subcutaneous tissue disorders) | 1
Rash, hands/feet (Skin and subcutaneous tissue disorders) | 1
redness areas under bunions (Skin and subcutaneous tissue disorders) | 1
abdominal pain (Gastrointestinal disorders) | 2
abdominal bloating (Gastrointestinal disorders) | 1
Anorexia (Gastrointestinal disorders) | 1
constipation (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 1
emesis (Gastrointestinal disorders) | 1
hematemesis (Gastrointestinal disorders) | 1
hemarrhoids (Gastrointestinal disorders) | 1
nausea (Gastrointestinal disorders) | 6
vomiting (Gastrointestinal disorders) | 2
asthenia (General disorders) | 1
malnourished (General disorders) | 1
pain-incision (General disorders) | 1
pain-both feet (General disorders) | 1
pain-post surgery (General disorders) | 1
throat sore (General disorders) | 1
mouth thrush (Infections and infestations) | 1
positive VRE/Enterococolis (Infections and infestations) | 1
elevated triglyceride (Metabolism and nutrition disorders) | 1
hyperglycemia (Metabolism and nutrition disorders) | 1
hypokalemia (Metabolism and nutrition disorders) | 2
hyponatremia (Metabolism and nutrition disorders) | 2
myalgia (Musculoskeletal and connective tissue disorders) | 1
right glenoid fossa fracture (Musculoskeletal and connective tissue disorders) | 1
shoulder pain (Musculoskeletal and connective tissue disorders) | 1
tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
bilateral lower extremities edema (Nervous system disorders) | 1
dizziness (Nervous system disorders) | 1
headache (Nervous system disorders) | 1
pain/tingling left arm (Nervous system disorders) | 1
somnolence (Nervous system disorders) | 1
tingling in feet (Nervous system disorders) | 1
altered mental status (Psychiatric disorders) | 1
confusion (Psychiatric disorders) | 1
difficulty concentrating (Psychiatric disorders) | 1
insomnia (Psychiatric disorders) | 2
dysuria (Renal and urinary disorders) | 1
urine incontinence (Renal and urinary disorders) | 1
urine pH less than 8 (Renal and urinary disorders) | 1
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
hiccups (Respiratory, thoracic and mediastinal disorders) | 1
productive cough (Respiratory, thoracic and mediastinal disorders) | 1
cough (Respiratory, thoracic and mediastinal disorders) | 4
wheezing (Respiratory, thoracic and mediastinal disorders) | 1
volume depletion (Vascular disorders) | 1
deep vein thrombosis, right upper extremity (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2
pedal edema (Blood and lymphatic system disorders) | 1
lower extremity edema (Blood and lymphatic system disorders) | 1

LIMITATIONS AND CAVEATS:
This study lost funding and was not able to enroll enough participants to do a complete review.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days